CLINICAL TRIAL: NCT01603017
Title: Nuclear Magnetic Resonance Therapy in Knee Osteoarthrosis: A Double Blind Ranomised Controlled Trial
Brief Title: Nuclear Magnetic Resonance Therapy in Knee Osteoarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Grampian (Other Government)
Responsible Party: Principal Investigator, S Barker, Consultant Orthopaedic Surgeon, NHS Grampian
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06/S0802/131
Record Dates: First submitted 2012-05-15; First posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthrosis
Keywords: Magnetic Resonance Therapy; Osteoarthrosis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo - no therapy (Placebo Comparator): Patients who were blinded but did not receive therapy
  Interventions: Device: MRI therapy (off)
- MRI therapy (Experimental): Patients receiving MRI therapy but blinded to it
  Interventions: Device: MRI therapy

INTERVENTIONS:
Device: MRI therapy — 5 treatments with magnetic field delivered to knee (n=50)
  Other Names: MBST-01, Version KSRT, Type 300 KSRT,; Serial Nos. 12100411 and 23490318,; manufactured by AD Elektronik GmbH, Wetzlar, Germany
  Arms: MRI therapy
Device: MRI therapy (off) — 5 treatment where MRI therapy machine was switched off (both patient and therapist blinded to this by use of electronic 'prescription cards'). (n=50)
  Other Names: MBST-01, Version KSRT, Type 300 KSRT,; Serial Nos. 12100411 and 23490318,; manufactured by AD Elektronik GmbH, Wetzlar, Germany
  Arms: Placebo - no therapy

SUMMARY:
Nuclear Magnetic Resonance Therapy (NMRT) is gaining as a novel mode of therapy in osteoarthrosis. A prospective double blind randomised study of 100 patients was conducted to investigate efficacy of NMRT in the treatment of mild to moderate osteoarthrosis (OA) of the knee joint.

The null hypothesis was that there is no benefit of NMRT over placebo in mild to moderate oteoarthosis of the knee.

DETAILED DESCRIPTION:
This study was approved by the Regional Ethics Committee. Patients were recruited from referrals made by General Practitioners to a single Orthopaedic Outpatient Department between October 2007 and February 2008. The study was a prospective placebo controlled, double blind randomised mono centric study with a follow up period of 6 months.

All potential trial participants demonstrated symptomatic mild to moderate OA of the knee joint diagnosed by an experienced consultant orthopaedic surgeon. Radiographic evidence was gathered by means of standard clinical standing antero-posterior and lateral radiographs of the knee.

Baseline assessment included :

1. clinical examination
2. active Range of movement
3. plain radiographs
4. WOMAC osteoarthritis index
5. Oxford Knee Score (OKS)
6. Severity of pain VAS.
7. Strength and frequency of any painkillers taken.
8. Phyasiotherapy Study design was directed at use of NMRT in a clinical setting. It was therefore considered valid to not restrict the use of the pain killers and physiotherapy. Positional Magnetic Resonance Imaging (pMRI) scan of the knee joint was undertaken.

Randomisation was carried out by means of visually identical computer chip cards numbered from 1 to 100 which had been independently programmed by the manufacturer. Thus, half of the computer chip cards (n=50) were programmed to activate the magnetic fields (= treatment group) and remaining half (n=50) were programmed not to activate magnetic fields (=placebo group) of the device. The research team and patients were blinded to the programmed activity of the cards. The magnetic resonance indicator LED lamp on the device was disabled by the manufacturer to ensure that the operator and patients were blinded to the therapy status. Every patient entering the study was asked to choose a numbered card from those available, and this card was then used to operate the device for that specific patient for all five sessions of NMRT.

The study used the manufacturer's clinical recommendation for therapy. Patients were subjected to one-hour sessions of NMRT (or placebo) on five consecutive days, giving a total of five hours of NMRT (or placebo). This was given on an outpatient basis.

The device is made up of twelve independently controlled coil systems that are spaced orthogonally. These are designed to produce a 3-dimensional therapy field. Along with a separately generated permanent magnetic field, the 3-dimensional therapy field forms a nuclear resonance field in the center of the coil system. The desired dose of NMRT is achieved with the help of MBST® - Treatment software, which is controlled by a computer chip card. The device can generate a magnetic field of 3.0 mT (typical) and maximum of 10 mT extending up to 30 cm around the device.

Patients were called for review at 1 week (1w), 1 month (1m), 3 months (3m) and 6 months (6m) when clinical examination, WOMAC osteoarthritis index and OKS were repeated. They were also asked to record VAS and details of painkillers taken during the week before each review. Due to the lack of recognised analgesia equivalencies, the quantity of pain killers taken were graded with reference to the amount and frequency taken at baseline - less than baseline was graded as 1, same as baseline was graded as 2 and more than baseline was graded as 3.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis of the knee(s)
* Moderately severe (grade 1-2)

Exclusion Criteria:

* Prior knee surgery
* Implanted metallic devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score | 12 weeks
  Patient administered validated questions

CONTACTS AND LOCATIONS:
Overall Officials: Simon L Barker, MD, Principal Investigator — NHS Grampian
Locations (1):
- Woodend Hospital, Aberdeen, Scotland, United Kingdom